CLINICAL TRIAL: NCT05789095
Title: Rate of Torque Development in Adolescents With Osgood-Schlatter: A Cross-sectional Case-control Study
Brief Title: Rate of Torque Development in Adolescents With Osgood-Schlatter
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kasper Krommes, Sensior Research Coordinator, PhD Fellow, Hvidovre University Hospital
Other Study IDs: H-20072873
Record Dates: First submitted 2023-02-23; First posted 2023-03-29 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Osgood-Schlatter Disease
Keywords: Adolescents; Rate of torque development; Osgood-Schlatter; Neuromuscular; Inhibition
MeSH Terms: conditions — Osteochondrosis; Inhibition, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case-group: 13 adolescents, 9-16 years, with Osgood-Schlatter Disease.
  Interventions: Other: Rate of torque development testing of knee flexors and knee extensors using a fixated handheld dynamometer (MicroFet 2, Hoggan, Scientific L.L.C., Salt Lake City, USA), sampling rate of 100hz)
- Control-group: 13 healthy adolescents, 9-16 years, without any knee pain, matched on age, sex and type of sport on the group-level.
  Interventions: Other: Rate of torque development testing of knee flexors and knee extensors using a fixated handheld dynamometer (MicroFet 2, Hoggan, Scientific L.L.C., Salt Lake City, USA), sampling rate of 100hz)

INTERVENTIONS:
Other: Rate of torque development testing of knee flexors and knee extensors using a fixated handheld dynamometer (MicroFet 2, Hoggan, Scientific L.L.C., Salt Lake City, USA), sampling rate of 100hz) — Participants and their parents/guardian receives information about the test procedures. Written informed consent is obtained before clinical examination and testing.
  Clinical testing is performed, anthropometric values are obtained and patient reported outcome measure is filled out, before the tests are performed. Cases will receive treatment for their condition and controls a movie ticket as compensation.

SUMMARY:
Osgood-Schlatter is a growth-related condition involving multiple different types of tissue in the tendon-bone interface at the tibial tubercle. Osgood-Schlatter affects one in ten adolescents causing persistent pain and reduced ability to maintain physical activities. Changes in rate of torque development is associated with decreased neuromuscular functioning and pain chronicity, thereby affecting athletic performances and general physical activities. However, changes in rate of torque development has not been investigate in patients with Osgood-Schlatter and could help characterize the condition and guide management.

The aim of the study is to investigate early and peak rate of torque development during maximal voluntary isometric knee extension and knee flexion in adolescents with Osgood-Schlatter, compared to a matched group of asymptomatic adolescents (controls), in a cross-sectional study.

The study will include 13 adolescent participants with Osgood-Schlatter and a group of 13 pain free controls matched on sex, age, and sports participation on the group level. Testing will include rate of torque measurements of knee extension and flexion for each limb with a fixated handheld dynamometer during a single test-session lasting approximately two hours. The examiner responsible for strength-testing will be blinded to case-status. Along with anthropometric data, participants will perform the anterior knee pain provocation test to assess pain-response to sustained knee loading, a countermovement jump test to assess power and jump height, and provide patient-reported measures of condition severity, pain, disability, and quality of life. Data collection will start March 2023 and is expected to finish by May 2023.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 9-16 years of age
* Presence of pain for 12 weeks or more
* Pain at tibial tubercle during loading activities
* Palpable pain at the tibial tuberosity

Exclusion Criteria:

* Previous knee or hip surgery
* Other main diagnose of anterior knee pain (patellofemoral pain, Sinding-Larsen Johansson disease, Jumpers knee, etc.)
* Hip and/or back pain interfering with activities of daily living or physical activities
* Suspicion of other main diagnose such as meniscal tears and or ligamental tears
* Unable to communicate verbally or orally in Danish

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents aged 9-16 residing in the uptake area of Copenhagen University Hospital, Amager-Hviodvre (1.8m total residents), who is made aware of the study be either 1) being referred to the orthopedic department for Osgood-Schlatter, 2) sees adverts and local sports clubs, or 3) sees the online advert on the research unit webpage
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of torque development (Nm/s/kg) at 0-200 ms during maximal isometric knee extension | Day 1
  Test performed seated on an examination bed with a belt-fixated handheld dynamometer (MicroFet 2, Hoggan Scientific, USA) at 60 degrees of knee flexion during a 5 second maximal exertion.
Rate of torque development (Nm/s/kg) at 0-100 ms during maximal isometric knee extension | Day 1
  Test performed seated on an examination bed with a belt-fixated handheld dynamometer (MicroFet 2, Hoggan Scientific, USA) at 60 degrees of knee flexion during a 5 second maximal exertion.
Peak rate of torque development (Nm/s/kg) during maximal isometric knee extension | Day 1
  Test performed seated on an examination bed with a belt-fixated handheld dynamometer (MicroFet 2, Hoggan Scientific, USA) at 60 degrees of knee flexion during a 5 second maximal exertion.
Time to peak force, during maximal isometric knee extension | Day 1
  Test performed seated on an examination bed with a belt-fixated handheld dynamometer (MicroFet 2, Hoggan Scientific, USA) at 60 degrees of knee flexion during a 5 second maximal exertion.
Rate of torque development (Nm/s/kg) at 0-200 ms during maximal isometric knee flexion | Day 1
  Test performed seated on an examination bed with a belt-fixated handheld dynamometer (MicroFet 2, Hoggan Scientific, USA) at 20 degrees of knee flexion during a 5 second maximal exertion.
Rate of torque development (Nm/s/kg) at 0-100 ms during maximal isometric knee flexion | Day 1
  Test performed seated on an examination bed with a belt-fixated handheld dynamometer (MicroFet 2, Hoggan Scientific, USA) at 20 degrees of knee flexion during a 5 second maximal exertion.
Peak rate of torque development (Nm/s/kg) during maximal isometric knee flexion | Day 1
  Test performed seated on an examination bed with a belt-fixated handheld dynamometer (MicroFet 2, Hoggan Scientific, USA) at 20 degrees of knee flexion during a 5 second maximal exertion.

SECONDARY OUTCOMES:
Pain during strength testing (NRS 10) | Day 1
  Numerical Pain Rating scale, 0-10 with 0 being no pain and 10 being worst imaginable.

OTHER OUTCOMES:
Knee osteoarthritis Outcome Score for children (KOOS Child) | Day 1
  The scale contains 7 questions answered through a 0-4 likert scale. The scale is normalized to a 0-100 score, with zero representing extreme knee problems and 100 representing no knee problems.
  In this study participants will fill out questions from the subscales "sport/rec", "quality of life" and question P1, P4, P6b and P6b from the "pain" subscale.
The Tampa Scale 17 (TSK-17) | Day 1
  The Tampa Scale is a 17-item questionnaire to evaluate fear avoidance behaviour in patients experiencing pain. It consists of two subscales on activity avoidance and somatic focus. The questions are rated on a 1-4 likert scale by the patient. The sum of the points are ranged from 17-68, with above 37 points being defined as "high level" of kinesiophobia.
Duration of pain | Day 1
  Participants self-reported duration of pain denoted in months
Worst pain in the last week | Day 1
  The perceived pain in the last week, rated on the Numerical Pain Rating scale, 0-10 with 0 being no pain and 10 being worst imaginable.
Worst pain in the last 24 hours | Day 1
  The perceived pain in the last 24 hours, rated on the Numerical Pain Rating scale, 0-10 with 0 being no pain and 10 being worst imaginable.
Current pain | Day 1
  The participants current pain on the Numerical Pain Rating scale, 0-10 with 0 being no pain and 10 being worst imaginable.
Counter Movement Jump Test | Day 1
  The participants will perform three trials of a countermovement jump which will be recorded on a smartphone camera (>240 frames per second). Subsequently, it will be analyzed for jump height using the MyJump 2 smartphone application.
Counter Movement Jump Test | Day 1
  The participants will perform three trials of a countermovement jump which will be recorded on a smartphone camera (>240 frames per second). Subsequently, it will be analyzed for power (W) using the MyJump 2 smartphone application.
Pain during Counter Movement Jump Test | Day 1
  The participants will perform three trials of a countermovement jump. The pain during each jump will be rated on the 0-10 Numerical Pain Rating scale, 0-10 with 0 being no pain and 10 being worst imaginable.
Anterior Knee Pain Provocation test | Day 1
  The participants will perform the Anterior Knee Pain Provocation test and rate the pain on the 0-10 Numerical Pain Rating Scale before and after the test. Only the affected knee is tested. For controls, the affected knee will be decided by coin toss.
Level of sports- participation and performance compared to before knee pain | Day 1
  Participants are asked if they perform either 1) at a higher level than before onset of knee pain, 2) at the same level as before onset of knee pain, or 3) at a lower level than before onset of knee pain
Level of physical activity compared to before knee pain | Day 1
  Participants are asked if they are either 1) more physically active than before onset of knee pain, 2) just as physically active as before onset of knee pain, or 3) are less physically active as before onset of knee pain

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be published either along the primary peer-reviewed journal publication if this will be available, otherwise to a public repository with a permanent Digital Object Identifier (DOI), for example, zenodo, figshare or similar.
Supporting Information: Study Protocol
Time Frame: The study protocol wil be uploaded to this registration once the study has been given an identifier from ClinicalTrials.gov
Access Criteria: No restrictions, but collaborators are required to adhere to the CC-BY-NC-ND 4.0 Licensing: Anyone can share this material, provided it remains unaltered in any way, this is not done for commercial purposes, and the original authors are credited and cited.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT05789095/Prot_SAP_000.pdf